CLINICAL TRIAL: NCT04036045
Title: Integrated Basis and Translational Approaches to Identify Early Biomarkers and Pathogenesis of Anthracycline Cardiotoxicity
Brief Title: Approaches to Identify Early Biomarkers and Pathogenesis of Anthracycline Cardiotoxicity
Status: Withdrawn | Type: Observational
Why Stopped: No funding, no participation
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 18-137
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Childhood Cancer
Keywords: Anthracycline induced cardiotoxicity
MeSH Terms: conditions — Neoplasms | interventions — Caves; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — pending
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cardiac MRI — Patients will have a cardiac MRI at four time points during the study
  Other Names: cMRI
Other: Echocardiogram — Patients will have an echocardiogram at four time points during the study
  Other Names: Echo
Other: Blood Draw — Patients will have blood drawn at four time points to analyze micro RNAs and Biomarkers before, during and after anthracycline treatment. Patients will also have one blood draw for future genetic sequencing.

SUMMARY:
Early microRNAs (miRs) and Cardiac Magnetic Resonance (CMR)-derived strain analysis and detection of genes contributing to Anthracycline-Induced Cardiotoxicity (AIC) sensitivity and resistance will identify pediatric cancer patients most and least likely to develop AIC.

DETAILED DESCRIPTION:
Plan is to enroll 110 children and adults (≥9 years old) newly diagnosed at CCMC and Nationwide Children's Hospital (55 per institution) who will receive anthracyclines as part of their chemotherapy regimen.

The duration of study participation will be approximately a year.

Patients will have a total of four study visits:

Baseline

1 week after patient's anthracycline cumulative dose hits between 60 and 100 mg/m2 After the patient has completed maximal therapy One year after completion of anthracycline treatments

Study tasks for all four visits will be:

Collection of clinical data Blood draw for micro RNA and Biomarkers Cardiac MRI Echocardiogram One time blood draw for genetics

ELIGIBILITY:
Inclusion Criteria:

* Age (≥ 9years old)
* Newly diagnosed with a malignancy that will receive ACs as part of their chemotherapy.
* Parental/caregiver consent and subject assent to enrollment.

Exclusion Criteria:

* Subject has contraindications to CMR.*
* Subject requiring sedation for CMR
* Subject too large to be safely accommodated by CMR
* Pregnancy tests are done routinely prior to chemotherapy, if test is positive the patient will be excluded
* Subject's serum creatinine above guidelines for adequate renal function. See table below:

Age (years) Male Female 6-10 1.0 mg/dL 1.0 mg/dL 10-13 1.2 mg/dL 1.2 mg/dL 13-16 1.5 mg/dL 1.4 mg/dL >16 1.7 mg/dL 1.4 mg/dL

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are > or equal to 9 years of age who are newly diagnosed with cancer who will receive anthracycline (s) as part of the their treatment regimen.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
CMR | From Baseline to one year after anthracycline therapy
  1. Increased myocardial T2 relaxation time in the myocardium compared to baseline as measured by T2 mapping technique

CONTACTS AND LOCATIONS:
Overall Officials: Olga Salazar, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Olga Salazar, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
Pending